CLINICAL TRIAL: NCT05742126
Title: A Randomized, Partial-Blind, Placebo and Positive-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Ascending Doses of HSK36273 in Healthy Subjects.
Brief Title: A Study of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Dosed of HSK36273 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HSK36273-101
Record Dates: First submitted 2022-11-09; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Healthy
Keywords: HSK36273; healthy; Phase I; continuous IV
MeSH Terms: interventions — Heparin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HSK36273 (Experimental): Multiple continuous IV infusion ascending doses in cohort 1-5
  Interventions: Drug: HSK36273
- Placebo (Placebo Comparator): 5 cohorts with matching placebo to HSK36273
  Interventions: Drug: Placebo
- Heparin sodium injection (Active Comparator): Cohort 1-2 with matching positive control to HSK36273
  Interventions: Drug: Heparin sodium injection

INTERVENTIONS:
Drug: HSK36273 — Multiple continuous IV infusion ascending doses for 5 days
  Arms: HSK36273
Drug: Placebo — Matching placebo
  Arms: Placebo
Drug: Heparin sodium injection — Matching positive control
  Arms: Heparin sodium injection

SUMMARY:
This is a single-center, Phase 1, placebo and positive-controlled, randomized, partial-blind, integrated, sequential ascending dose / multiple ascending dose study.The safety, tolerability, pharmacokinetics and pharmacodynamics of multiple continuous IV infusion ascending doses of HSK36273 in healthy volunteers will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females, 18 to 45 years of age (inclusive) at Screening.
2. Body Mass Index (BMI) ≥ 18.0 and ≤ 28.0 kg/m2 and a weight of at least 45 kg for female and 50 kg for male.
3. The subject must be willing and able to provide written informed consent
4. Medically healthy without clinically significant abnormalities at Screening and predose on Day 1, including:

   1. Physical examination without any clinically relevant findings.
   2. Three conventional 12-ECG recordings (the average of the three measurements will be used to determine eligibility) were consistent with normal cardiac conduction and function.
   3. QT interval corrected using the Fridericia method (QTcF) between 350 to 450 msec for male subjects and 350 to 470 msec for female subjects, inclusive.
   4. Normal laboratory tests (hematology, biochemistry, urinalysis, coagulation tests (aPTT and PT).
   5. No clinically significant findings in serum chemistry, hematology, coagulation, and urinalysis tests as deemed by the Investigator.
5. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
6. Willing and able to comply with all study evaluations and adhere to protocol schedules and constraints.

Exclusion Criteria:

1. History or presence of major diseases of the cardiovascular, respiratory, digestive, urological, hematologic, endocrine, immunologic, skin or nervous system, as well as any acute illness or surgical procedure within the past 3 months as determined by the investigator to be clinically relevant.
2. History of abnormal bleeding episodes, e.g. nosebleeds, or abnormally heavy periods, or extensive bleeding after injury, surgery or dental work within 3 months prior to screening.
3. Any clinically Laboratory tests during the screening period were abnormal and clinically significant as judged by the investigator. Liver function test results (i.e., aspartate aminotransferase [AST], alanine aminotransferase [ALT], and gamma glutamyl transferase[GGT]) and total bilirubin elevated above the ULN.
4. Positive test results for active HIV, hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibodies (Abs).
5. Hemoglobin or hematocrit clinically significantly less than lower limits of normal at screening.
6. History of drug abuse in the 12 months prior to the first administration of the study drug or alcohol abuse in the 3 months prior.
7. A clinically significant allergic reaction that the investigator believes interferes with the subject's ability to participate in the trial; Known allergies to any of the study drug ingredients, allergy to anticoagulants or antiplatelet drugs or obvious adverse reactions, allergic to two or more drugs or food, allergic to any ingredient in this product and auxiliary materials.
8. Donate blood or plasma within 3 months prior to the first administration of the study drug, or lose more than 400mL of whole blood, or receive blood transfusion within 1 year prior to the first administration of the study drug.
9. History of Participating in another investigational clinical trial within 90 days before the first administration of the study drug.
10. Poor venous access that would hamper a 5-day infusion.
11. Positive pregnancy test at screening or check-in (Day -1).
12. Participation in a clinical trial involving the administration of an investigational or marketed drug within 30 days (90 days for biologics), or five (5) half-lives, whichever is longer, prior to the first dosing or concomitant participation in an investigational study involving no drug administration.
13. Any other factors considered by the investigator to be inappropriate for participation in the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
The number and severity of treatment emergent adverse events (TEAEs) . | Day1 to Day8
  To assess the safety and tolerability of multiple of HSK36273 following 24-hour continuous IV infusions administered over 5 consecutive days with ascending doses in healthy subjects

SECONDARY OUTCOMES:
AUC0-24h | within 1 hour before administration until 24 hours after starting administration
  Area under the drug concentration-time curve, from time 0h to 24h
AUC0-144h | within 1 hour before administration until 144 hours after administration
  Area under the drug concentration-time curve, from time 0h to 144h
Css | within 1 hour before administration until 144 hours after administration
  Steady-State Concentration with a the Initiation of Continuous IV 5-day Infusion of HSK36273
Tss | within 1 hour before administration until 144 hours after administration
  Time to Reach a Steady-State Concentration Following a the Initiation of Continuous IV 5-day Infusion of HSK36273
t1/2 | 24 hours after administration
  Apparent terminal half-life
CL | 24 hours after administration
  Apparent total clearance of drug
Vd | 24 hours after administration
  Apparent volume of distribution
Activated Partial Thromboplastin Time (aPTT) | within 1 hour before administration until 144 hours after administration
  Clotting Biomarker Activated Partial Thromboplastin Time During the Course of a Continuous IV 5-day Infusion of HSK36273
Prothrombin Time (PT) | within 1 hour before administration until 144 hours after administration
  Clotting Biomarker Prothrombin During the Course of a Continuous IV 5-day Infusion of HSK36273
Activated Clotting Time (ACT) | within 1 hour before administration until 144 hours after administration
  Clotting Biomarker Activated Clotting Time During the Course of a Continuous IV 5-day Infusion of HSK36273
FXIa | within 1 hour before administration until 144 hours after administration
  Change from baseline in factor XI activity

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China